CLINICAL TRIAL: NCT03901820
Title: Evaluation of a Drug Interactions Software to Limit Polypharmacy (Evaluación de un Programa de Interacciones Medicamentosas Para Limitar la Polifarmacia)
Brief Title: Evaluation of a Drug Interactions Software to Limit Polypharmacy
Acronym: SIMDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Guillermo Alberto Keller, Head of Pharmacovigilance Program, University of Buenos Aires
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RB-001
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Polypharmacy; Elderly; Inpatient; Drug Interaction
Keywords: Electronic Record; Drug interaction; Polypharmacy; Elderly; Adverse Drug reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: An electronic medical record, DrApp, will be used, which will include a drug interaction program, SIMDA, which will automatically indicate the medication prescriptions that involve a risk for the patient.
  The first indication of each patient admitted to two rooms of the Internal Medicine Department of the Hospital de Clínicas José de San Martín will be registered. The indications will be compared in the 4 months prior to the incorporation of the SIMDA program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum number of patients that will be included in each stage is 100.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DrApp Without SIMDA (No Intervention): There are approximately 100 inpatients in whom the indications were registered through the use of DrApp, before the implementation of the drug interactions detection module.
- DrApp With SIMDA (Experimental): There are approximately 100 inpatients in whom the indications were registered through the use of DrApp, AFTER the implementation of the drug interactions detection module (SIMDA).
  Interventions: Device: Medication Interaction System of Dr App (SIMDA)

INTERVENTIONS:
Device: Medication Interaction System of Dr App (SIMDA) — A module for the electronic clinical records allowing detection of the potential drug interactions
  Other Names: SIMDA
  Arms: DrApp With SIMDA

SUMMARY:
Multiple morbidity is increasing, especially in elderly people, with a corresponding increase in polypharmacy and inappropriate prescriptions. According to different evaluations, between 25 and 75% of patients aged 75 or older are exposed to 5 or more drugs. There is increasing evidence that polypharmacy can cause more harm than good, especially in elderly people, due to factors such as drug-drug and drug-disease interactions.

Many strategies were proposed to reduce polypharmacy and inappropriate prescribing, but there is little evidence to show benefit. There is an urgent need to implement effective strategies. The application methodology must be simple so that it does not fail in daily practice.

For the current plan, an electronic medical record, named "DrApp", will be used, which will include a drug interaction program, SIMDA, which will automatically indicate the medication prescriptions that involve a risk for the patient.

The first indication of each patient admitted to two rooms of the Internal Medicine Department of the Hospital de Clínicas José de San Martín will be registered. The indications will be compared in the 4 months prior to the incorporation of the SIMDA program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum number of patients that will be included in each stage is 100.

The primary end point is to compare the total number of indications per inpatient, before the availability of the SIMDA program and after the application of this program.

The objective is to evaluate if the computer program of detection of drug interactions allows to limit the polypharmacy in hospitalized patients.

DETAILED DESCRIPTION:
Multiple morbidity is increasing, especially in elderly people, with a corresponding increase in polypharmacy and inappropriate prescriptions. According to different evaluations, between 25 and 75% of patients aged 75 or older are exposed to 5 or more drugs. There is increasing evidence that polypharmacy can cause more harm than good, especially in elderly people, due to factors such as drug-drug and drug-disease interactions.

Many strategies were proposed to reduce polypharmacy and inappropriate prescribing, but there is little evidence to show benefit. There is an urgent need to implement effective strategies. The application methodology must be simple so that it does not fail in daily practice.

For the current plan, an electronic medical record, named "DrApp", will be used, which will include a drug interaction program, SIMDA, which will automatically indicate the medication prescriptions that involve a risk for the patient.

The first indication of each patient admitted to two rooms of the Internal Medicine Department of the Hospital de Clínicas José de San Martín will be registered. The indications will be compared in the 4 months prior to the incorporation of the SIMDA program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum number of patients that will be included in each stage is 100.

The primary end point is to compare the total number of indications per inpatient, before the availability of the SIMDA program and after the application of this program.

The objective is to evaluate if the computer program of detection of drug interactions allows to limit the polypharmacy in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients interned in the medical clinic room of the Hospital de Clínicas José de San Martín

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of polypharmacy cases detected in two internal medicine hospitalization units of a University Hospital | 1 year
  Through the electronic medical record called DrApp, the quantity of medicines prescribed to each patient is quantified and used for calculation of polypharmacy prevalence in tha basal period (pre-introduction of SIMDA) and late period (Post introduction of SIMDA).

SECONDARY OUTCOMES:
SIMDA associated change in the number of total prescribed drug per patient | 1 year
  Change in total prescribed drug per patient will be calculated as the differene between basal total prescribed drug per patient (Pre-SIMDA) minus resulting total prescribed drug per patient (Post-SIMDA)
Number of total drug interactions per patient and subclassification by severity (in post-SIMDA period). | 1 year
  The addition of the application called SIMDA, will allow detecting the presence of drug interactions and their severity in the second phase. These will be reported as the total number of interactions reported per patient, and subclassificated into number of mild (no need to take action), moderate (require patient monitoring), and severe (possible contraindication) interactions detected per patient.
difference between Number of total drug interactions per patient in the local environment with those reported in the literature at the international level | 1 year
  The difference will be calculated as the number of total drug interactions per patient minus the value (number of drug interaction per patient) reported in the bibliography at international level in similar populations.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Barcia, MD, Principal Investigator — Universidad de Buenos Aires, Hospital de Clínicas José de San Martín; Francisco Azzato, MD PhD, Study Director — Universidad de Buenos Aires, Hospital de Clínicas José de San Martín; Roberto A Diez, MD PhD, Study Director — Universidad de Buenos Aires, Facultad de Medicina, Centro de Vigilancia y Seguridad de Medicamentos; Guillermo A Keller, MD PhD, Principal Investigator — Universidad de Buenos Aires, Facultad de Medicina, Centro de Vigilancia y Seguridad de Medicamentos
Locations (1):
- Hospital de Clínicas José de San Martín, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
There is an intention to publish all the results obtained and share them with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year after study termination

REFERENCES:
- [Background] Sonnichsen A, Trampisch US, Rieckert A, Piccoliori G, Vogele A, Flamm M, Johansson T, Esmail A, Reeves D, Loffler C, Hock J, Klaassen-Mielke R, Trampisch HJ, Kunnamo I. Polypharmacy in chronic diseases-Reduction of Inappropriate Medication and Adverse drug events in older populations by electronic Decision Support (PRIMA-eDS): study protocol for a randomized controlled trial. Trials. 2016 Jan 29;17:57. doi: 10.1186/s13063-016-1177-8. PMID 26822311
- [Background] Rieckert A, Sommerauer C, Krumeich A, Sonnichsen A. Reduction of inappropriate medication in older populations by electronic decision support (the PRIMA-eDS study): a qualitative study of practical implementation in primary care. BMC Fam Pract. 2018 Jul 9;19(1):110. doi: 10.1186/s12875-018-0789-3. PMID 29986668
- [Background] Clyne B, Bradley MC, Hughes CM, Clear D, McDonnell R, Williams D, Fahey T, Smith SM; OPTI-SCRIPT study team. Addressing potentially inappropriate prescribing in older patients: development and pilot study of an intervention in primary care (the OPTI-SCRIPT study). BMC Health Serv Res. 2013 Aug 14;13:307. doi: 10.1186/1472-6963-13-307. PMID 23941110
- [Background] Clyne B, Cooper JA, Hughes CM, Fahey T, Smith SM; OPTI-SCRIPT study team. A process evaluation of a cluster randomised trial to reduce potentially inappropriate prescribing in older people in primary care (OPTI-SCRIPT study). Trials. 2016 Aug 3;17(1):386. doi: 10.1186/s13063-016-1513-z. PMID 27488272
- [Background] Bril F, Castro V, Centurion IG, Espinosa J, Keller GA, Gonzalez CD, Riera MC, Saubidet CL, Di Girolamo G, Pujol GS, Alvarez PA. A Systematic Approach to Assess the Burden of Drug Interactions in Adult Kidney Transplant Patients. Curr Drug Saf. 2016;11(2):156-63. doi: 10.2174/157488631102160429003742. PMID 27194037
- [Background] Alvarez PA, Bril F, Castro V, Meiville I, Gonzalez CD, Centurion IG, Parejas G, Riera CS, Saubidet CL, Di Girolamo G, Keller GA. Adverse drug reactions as a reason for admission to an internal medicine ward in Argentina. Int J Risk Saf Med. 2013;25(3):185-92. doi: 10.3233/JRS-130596. PMID 24047689
- [Derived] Barcia RE, Keller GA, Azzato F, Diez RA, Sielecki M, Kleine RS, Lescano JA, Giunti G. Development and Implementation of the Hdc.DrApp.la and SIMDA Programs to Reduce Polypharmacy and Drug-drug Interactions in Patients Hospitalized in Internal Medicine. Rev Recent Clin Trials. 2023;18(2):156-166. doi: 10.2174/1574887118666230208124744. PMID 36752290